CLINICAL TRIAL: NCT01837251
Title: A Prospective Randomized Phase III Trial of Carboplatin/Gemcitabine/Bevacizumab vs. Carboplatin/Pegylated Liposomal Doxorubicin/Bevacizumab in Patients With Platinum-sensitive Recurrent Ovarian Cancer
Brief Title: Evaluation of Optimal Treatment With Bevacizumab in Patients With Platinum-sensitive Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AGO Research GmbH (Industry)
Collaborators: Arbeitsgemeinschaft Gynaekologische Onkologie Austria (Other); ARCAGY/ GINECO GROUP (Other); Australia New Zealand Gynaecological Oncology Group (Other); Scottish Gynaecological Cancer Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OVAR 2.21 / ENGOT ov-18
Record Dates: First submitted 2013-04-16; First posted 2013-04-23 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Recurrent Platinum-sensitive Ovarian Cancer
Keywords: Ovarian Carcinoma; Bevacizumab; Gemcitabine; PLD; pegylated liposomal doxorubicin; Carboplatin; best therapeutic index; progression-free survival
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; 1-dodecylpyridoxal; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (No Intervention): Patients receive bevacizumab 15 mg/kg iv on day 1 followed by gemcitabine 1000mg/m² iv on day 1 & 8 and carboplatin AUC4 iv on day 1 every 3 weeks for up to 6 cycles in the absence of progression disease or unacceptable toxicities. Patients then continue to receive bevacizumab 15 mg/kg iv every 3 weeks until progression disease or unacceptable toxicities.
- Research Arm (Experimental): Patients receive bevacizumab 10 mg/kg iv on day 1 & 15 followed by PLD 30mg/m² iv on day 1 carboplatin AUC4 iv on day 1 every 4 weeks for up to 6 cycles in the absence of progression disease or unacceptable toxicities. Patients then continue to receive bevacizumab 15 mg/kg iv every 3 weeks until progression disease or unacceptable toxicities.
  Interventions: Drug: Carboplatin; Drug: PLD; Biological: Bevacizumab

INTERVENTIONS:
Drug: Carboplatin
  Arms: Research Arm
Drug: PLD
  Arms: Research Arm
Biological: Bevacizumab
  Arms: Research Arm

SUMMARY:
Evaluation of the best therapeutic index for patients with platinum-sensitive ovarian cancer when treatment with bevacizumab and gemcitabine/carboplatin or with bevacizumab and PLD/carboplatin.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of epithelial ovarian carcinoma or fallopian tube carcinoma or primary peritoneal carcinoma
2. First disease recurrence >6 months after first-line platinum-based chemotherapy
3. Patients with measurable or non-measurable disease (RECIST v1.1) or CA 125 assessable disease (GCIG criteria) or histological proven diagnosis of relapse
4. In case of cytoreductive surgery for recurrence, patients must be able to commence cytotoxic chemo-therapy within 8 weeks after cytoreductive surgery
5. ECOG PS 0-2
6. Absolute Neutrophil Count >= 1.5 x 10^9/L; Platelets >= 100 x 10^9/L; Hemoglobin >= 9.5 g/dL
7. Patients not receiving anticoagulant medication who have an International Normalized Ratio <= 1.5 and an Activated ProThrombin Time <= 1.5 x ULN
8. Serum bilirubin <= 2 x ULN; Serum transaminases <= 2.5 x ULN (<= 5 x ULN in the presence of liver metastasis)
9. Serum creatinine < 1.6 mg/dL or creatinine clearance >= 40 mL/min; Glomerular filtration rate > 40 ml/min (estimates based on the Cockroft-Gault or Jelliffe formula); Urine dipstick for proteinuria < 2+. If urine dipstick is >= 2+, 24 hour urine collection must demonstrate <= 1 g of protein in 24 hours
10. Normal blood pressure or adequately treated and controlled hypertension (either systolic BP ≤ 140 mmHg and/or diastolic BP ≤ 90 mmHg)

Exclusion Criteria:

1. Ovarian tumors of low malignant potential
2. Malignancies other than ovarian cancer within 5 years prior to randomization
3. Administration of other simultaneous chemotherapy drugs, any other anticancer therapy or anti-neoplastic hormonal therapy, or simultaneous radiotherapy during the trial treatment period
4. Any previous radiotherapy to the abdomen or pelvis
5. Known hypersensitivity to used chemotherapeutic agents in this trial and bevacizumab and its excipients, chinese hamster ovary cell products or other recombinant human or humanised antibodies
6. Current or recent chronic use of aspirin > 325 mg/day
7. Surgery (including open biopsy) within 4 weeks prior to anticipated first dose of Bevacizumab
8. History of VEGF therapy related abdominal fistula or gastrointestinal perforation
9. Current, clinically relevant bowel obstruction, including sub-occlusive disease, related to underlying disease
10. Patients with evidence of abdominal free air not explained by paracentesis or recent surgical procedure
11. Previous Cerebro-Vascular Accident , Transient Ischaemic Attack or Sub-Arachnoid Haemorrhage
12. Prior history of hypertensive crisis or hypertensive encephalopathy
13. Clinically significant disease, including: myocardial infarction or unstable angina within ≤ 6 months of randomization; New York Heart Association (NYHA) >= grade 2 Congestive Heart Failure; poorly controlled cardiac arrhythmia despite medication; peripheral vascular disease grade >= 3
14. LVEF defined by ECHO/MUGA below the institutional lower limit of normal
15. Significant traumatic injury during 4 weeks prior to randomization
16. Current brain metastases or spinal cord compression
17. History or evidence upon neurological examination of central nervous system disease
18. Non-healing wound, active ulcer or bone fracture
19. History or evidence of thrombotic or hemorrhagic disorders within 6 months prior to randomization
20. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic coagulation)
21. Fertile woman of childbearing potential not willing to use adequate contraception (oral contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) for the duration of the trial and at least 6 months afterwards
22. Pregnant or lactating women
23. Requirement of therapeutic anticoagulation using marcumar, warfarin or PTT-prolonging heparin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
investigator-determined progression-free survival | every 12 weeks until progression or up to 30 months (whichever occurs first)

SECONDARY OUTCOMES:
biological progression-free survival by serum CA 125 | every 3 weeks until progression or up to 30 months (whichever occurs first)
Health related Quality of Life (QoL) | Baseline and then every 12 weeks until investigator-determined progresssion-free survival and thereafter at every visit for th 5-years follow-up or death (whichever occurs first)
Safety and Tolerability, i.e. type, frequency, severity and duration o adverse reactions | every 3 weeks, 30 months after start of treatment or if applicable 4 weeks after last dose of bevacizumab (whichever occurs later)
Overall Survival | every 3 weeks during treatment with bevacizumab, thereafter every 6 months; for up 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacobus Pfisterer, PhD MD, Study Chair — AGO Study Group
Locations (193):
- Australia (19):
  - Bankstown-Lidcombe Hospital, Bankstown
  - Chris O'Brien Lifehouse, Camperdown
  - NCCI - Coffs Harbour Hospital, Coffs Harbour
  - The Townsville Hospital, Douglas
  - Peninsula Health - Frankston Hospital, Frankston
  - Andrew Love Cancer Centre Geelong, Geelong
  - Royal Brisbane & Women's Hospital, Herston
  - Royal Hobart Hospital, Hobart
  - St. George Hospital, Kogarah
  - ICON Cancer Care Centre, Milton
  - Nambour General Hospital, Nambour
  - Sir Charles Gairdner, Nedlands
  - North Coast Cancer Institute, Port Macquarie
  - Royal Hospital for Women, Randwick
  - Mater Adult Hospital, South Brisbane
  - Gold Coast University Hospital, Southport
  - Royal North Shore Hospital, St Leonards
  - St. John of God Hospital, Subiaco
  - Border Medical Oncology, Wodonga
- Austria (6):
  - MUG-Universitätsklinik für Frauenheilkunde Graz, Graz
  - MUI-Universität für Frauenheilkunde, Innsbruck
  - AKH Linz, Linz
  - BHS Linz, Linz
  - SALK-LKH Salzburg, Universitätsklinik für Frauenheilkunde und Geburtshilfe, Salzburg
  - MUW-AKH Wien, Vienna
- UZ Leuven, Leuven, Belgium
- France (42):
  - ICO Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de Blois, Blois
  - Clinique Tivoli, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Centre Hospitalier de Cholet, Cholet
  - Hôpital Antoine Béclère, Clamart
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier la Dracénie, Draguignan
  - Centre Hospitalier Général de Gap, Gap
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Hôpital Michallon, Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - Institut d'Oncologie Hartmann, Levallois-Perret
  - Centre Oscar Lambret, Lille
  - Hôpital Privé Clairval, Marseille
  - Institute Paoli Clamettes, Marseille
  - Hôpital Mercy, Metz
  - Hôpital de Mont-de-Marsan, Mont-de-Marsan
  - ICM Val d'Aurelle, Montpellier
  - Hôpital Emile Muller, Mulhouse
  - Centre d'Oncologie de Gentilly, Nancy
  - Centre Catherine de Sienne, Nantes
  - Centre Hospitalier Régional d'Orleans, Orléans
  - Group Hospitalier Saint-Joseph, Paris
  - Centre Catalan d'Oncologie, Perpignan
  - Clinique Francheville, Périgueux
  - Centre Eugène Marquis, Rennes
  - HôpitauxDrôme Nord - Site de Ramons, Romans-sur-Isère
  - Centre Henri Becquerel, Rouen
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - ICO Centre René Gauducheau, Saint-Herblain
  - Clinique Mutualiste de l'Estuaire, Cité Sanitaire, Saint-Nazaire
  - Centre Paul Strauss, Strasbourg
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Centre Hospitalier de Thonon-les-Bains, Thonon-les-Bains
  - Clinique Pasteur, Toulouse
  - Clinique Saint Jean du Languedoc, Toulouse
  - Centre Hospitalier Bretagne Atlantique, Vannes
  - Hôpital Privé Villeneuve d'Ascq, Institut de Canérologie, Villeneuve-d'Ascq
- Germany (121):
  - Kreisklinik Altötting-Burghausen, Altötting
  - Klinikum St. Marien, Amberg
  - Klinikum Aschaffenburg, Aschaffenburg
  - Klinikum Augsburg, Augsburg
  - Hochtaunus-Klinik, Bad Homburg
  - Charité - Universitätsmedizin Berlin, Berlin
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Praxisklinik Krebsheilkunde für Frauen, Berlin
  - Augusta-Kranken-Anstalt Bochum, Bochum
  - Johanniter-Krankenhaus, Bonn
  - Medizinisches Zentrum Bonn-Friedensplatz, Bonn
  - Schwerpunktpraxis für Onkologie / Hämatologie, Bottrop
  - Städtisches Klinikum Brandenburg, Brandenburg
  - Gynäkologisch-Onkologische Gemeinschaftspraxis, Braunschweig
  - DIAKO Ev. Diakonie-Krankenhaus, Bremen
  - Gynaekologicum Bremen, Bremen
  - Klinikum Bremen-Mitte, Bremen
  - Klinikum Chemnitz, Chemnitz
  - St. Elisabeth-Krankenhaus Hohenlind, Cologne
  - Universitätsklinikum Köln, Cologne
  - Klinikum Darmstadt, Darmstadt
  - Donau-Isar-Kliniken, Klinikum Deggendorf, Deggendorf
  - Städtisches Klinikum Dessau, Dessau
  - Klinikum Dortmund, Dortmund
  - Onkozentrum Dresden, Dresden
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Kaiserswerther Diakonie, Florence-Nightingale-Krankenhaus, Düsseldorf
  - Universitätsfrauenklinik Düsseldorf, Düsseldorf
  - Rottal-Inn-Klinik Eggenfelden, Eggenfelden
  - Universitätsklinikum Erlangen, Erlangen
  - Klinikum Essen Mitte, Essen
  - Universitätsklinikum Essen, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - DIAKO Flensburg, Flensburg
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Klinikum Frankfurt Höchst, Frankfurt
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsfrauenklinik Freiburg, Freiburg im Breisgau
  - Kreiskrankenhaus Freudenstadt, Freudenstadt
  - Klinikum Fürth, Fürth
  - Franziskus-Hospital Harderberg, Georgsmarienhütte
  - HELIOS-Klinikum Gifhorn, Gifhorn
  - Onkologische Kooperation Harz, Goslar
  - Die Frauenarztpraxis in Grafing, Grafing
  - Universitätsmedizin Greifswald, Greifswald
  - Universitätsklinikum Halle, Halle
  - Albertinen Krankenhaus, Hamburg
  - Marienkrankenhaus Hamburg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Sana-Klinikum Hameln-Pyrmont, Hamelin
  - Klinikum Hanau, Hanau
  - Friederikenstift, Hanover
  - Gynäkologisch-Onkologische Praxis Hannover, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Paracelsus-Klinik, Henstedt-Ulzburg
  - Praxis Dres. Uleer / Pourfard, Hildesheim
  - Klinikum Itzehoe, Itzehoe
  - Universitätsklinikum Jena, Jena
  - St. Vincentius Kliniken, Karlsruhe
  - Klinikum Kassel, Kassel
  - Klinikum Kempten, Kempten
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Zentrum für Gynäkologische Onkologie, Kiel
  - Klinikum Konstanz, Konstanz
  - Klinikum Kulmbach, Kulmbach
  - Asklepios Klinik Lich, Lich
  - St. Vincenz Krankenhaus, Limburg
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Onkologische Schwerpunktpraxis Lüneburg, Lüneburg
  - Klinik St. Marienstift, Magdeburg
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsmedizin Mainz, Mainz
  - Universitätsfrauenklinik Mannheim, Mannheim
  - Universitätsklinikum Gießen und Marburg, Marburg
  - Johannes Wesling Klinikum, Minden
  - Klinikum rechts der Isar, München
  - LMU München, Frauenklinik Großhadern, München
  - Rotkreuzklinikum München, München
  - Universitätsklinikum Münster, Münster
  - Kliniken des Landkreises Neumarkt, Neumarkt
  - Lukaskrankenhaus, Neuss
  - MVZ Nordhausen, Nordhausen
  - Klinikum Nürnberg, Nuremberg
  - Klinikum Offenbach, Offenbach
  - Ortenau-Klinikum, Offenburg
  - Marienhospital, Osnabrück
  - St. Vincenz Krankenhaus, Paderborn
  - Onkologische Praxis Pinneberg, Pinneberg
  - Harzklinikum Quedlinburg, Quedlinburg
  - Onkologie Ravensburg, Ravensburg
  - imland Klinik Rendsburg, Rendsburg
  - Klinikum am Steinenberg, Reutlingen
  - Universitätsfrauenklinik Rostock, Rostock
  - Thüringen-Kliniken, Saalfeld
  - Caritasklinikum St. Theresia, Saarbrücken
  - Praxis Dr. med. W. Dietz, Salzgitter
  - Diakonie-Klinikum Schwäbisch Hall, Schwäbisch Hall
  - Leopoldina-Krankenhaus, Schweinfurt
  - HELIOS Kliniken Schwerin, Schwerin
  - Diakonie Klinikum Jung-Stilling, Siegen
  - Klinikum Schaumburg, Krankenhaus Stadthagen, Stadthagen
  - Klinikum Starnberg, Starnberg
  - g.Sund Gyn. Kompetenzzentrum, Stralsund
  - Marienhospital Stuttgart, Stuttgart
  - Robert-Bosch-Krankenhaus, Stuttgart
  - SRH Zentralklinikum Suhl, Suhl
  - Kreiskrankenhaus "J. Kentmann", Torgau
  - Klinikum Traunstein, Traunstein
  - Klinikum Mutterhaus, Trier
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsfrauenklinik Ulm, Ulm
  - Praxis Dr. med. W. W. Reiter, Viersen
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen, Villingen-Schwenningen
  - Lahn-Dill-Kliniken Wetzlar, Wetzlar
  - Dr. Horst Schmidt Kliniken, Wiesbaden
  - St. Josefs Hospital Wiesbaden, Wiesbaden
  - amO am Klieversberg, Wolfsburg
  - Klinikum Worms, Worms
  - Heinrich-Braun-Klinikum, Zwickau
- United Kingdom (4):
  - Gwynedd Hospital, Bangor
  - Velindre Cancer Centre, Cardiff
  - The Beatson West of Scotland Cancer Center, Glasgow
  - Glan Clywd Hospital, Rhyl

REFERENCES:
- [Result] Pfisterer J, Shannon CM, Baumann K, Rau J, Harter P, Joly F, Sehouli J, Canzler U, Schmalfeldt B, Dean AP, Hein A, Zeimet AG, Hanker LC, Petit T, Marme F, El-Balat A, Glasspool R, de Gregorio N, Mahner S, Meniawy TM, Park-Simon TW, Mouret-Reynier MA, Costan C, Meier W, Reinthaller A, Goh JC, L'Haridon T, Baron Hay S, Kommoss S, du Bois A, Kurtz JE; AGO-OVAR 2.21/ENGOT-ov 18 Investigators. Bevacizumab and platinum-based combinations for recurrent ovarian cancer: a randomised, open-label, phase 3 trial. Lancet Oncol. 2020 May;21(5):699-709. doi: 10.1016/S1470-2045(20)30142-X. Epub 2020 Apr 16. PMID 32305099
- See also: Homepage of AGO Study Group — http://www.ago-ovar.de